CLINICAL TRIAL: NCT07212998
Title: Plasma Resuscitation Early for Evaluating Volume and Endotheliopathy of Thermal Injury (PREEVEnT) Trial
Acronym: PREEVEnT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jason Sperry (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Jason Sperry, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY25030138; HT9425-24-3-0002 (Other Grant/Funding Number: U.S. Department of Defense (DoD))
Record Dates: First submitted 2025-07-31; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Burn Injury; Thermal Burn
Keywords: burn; plasma resuscitation
MeSH Terms: conditions — Burns | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: permuted block design with variable block sizes of 4 and 6, stratified by site
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Plasma Resuscitation (Experimental): Subjects will receive early plasma resuscitation initiated in the emergency department/burn resuscitation area over an approximate 4-hour period from the time of randomization, stratified by Total Body Surface Area (TBSA)%.
  Interventions: Biological: Plasma
- Standard Care (Active Comparator): Subjects will receive resuscitation following individual site standard burn resuscitation practice.
  Interventions: Biological: Standard care

INTERVENTIONS:
Biological: Plasma — urgent release early plasma resuscitation following burn/thermal injury
  Arms: Early Plasma Resuscitation
Biological: Standard care — Standard resuscitation as dictated by institutional protocol
  Arms: Standard Care

SUMMARY:
The Plasma Resuscitation Early for Evaluating Volume and Endotheliopathy of Thermal Injury (PREEVEnT) trial will be a 6-year (4-year enrollment), open label, phase-3, multi-center, early in-hospital phase randomized trial utilizing burn centers from within the LITES network and will enroll approximately 750 injured adult patients who have suffered large 2nd or 3rd degree thermal burns on at least 20% of their body surface requiring burn resusciation. The objective is to determine if initiating plasma resuscitation as soon as possible upon arrival to an emergency department or burn unit is the most effective resuscitation for those who have experienced large thermal burns and significantly reduces the morbidity and mortality attributable to post-injury complications as compared to standard in-hospital resuscitation practice.

ELIGIBILITY:
Inclusion Criteria:

* Estimated ≥ 20% Total Body Surface Area burn/thermal injury with 2nd or 3rd degree depth
* Anticipated admission to burn ICU

Exclusion Criteria:

* Estimated rBaux score <55
* Not expected to survive >24 hours
* Wearing NO PREEVENT opt-out bracelet
* Age > 75 or < 18 years of age
* Concomitant traumatic injury with hemorrhagic shock
* Isolated chemical burn/injury
* Isolated deep electrical burn/injury
* Known prisoner
* Known pregnancy
* Cardiac arrest with > 5 continuous minutes of CPR
* Concern for anoxic injury/ fixed pupils bilaterally
* Objection to study voiced by subject or family member at the scene or at the emergency department/burn center

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2030-04 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
28-day Mortality or Persistent Organ Dysfunction | 28 days
  Composite outcome consisting of 28-day all-cause mortality, or 28-day Persistent Organ Dysfunction (POD) requiring support defined as 1) any intravenous vasopressor requirement, or 2) any renal replace therapy, or 3) any ventilator support/mechanical ventilation, or 4) continued need for intensive care unit (ICU) admission at 28 days.

SECONDARY OUTCOMES:
14-day mortality or Persistent Organ Dysfunction | 14 days
  Composite Outcome consisting of of 14-day all-cause mortality, or 14-day Persistent Organ Dysfunction requiring support (any intravenous vasopressor requirement, or any renal replace therapy, or any ventilator support, or continued need for intensive care unit (ICU) admission at 14 days)
Arterial or venous thromboembolism in first 7 days | 7 days
  Pulmonary embolism, venous thrombosis, or arterial thrombosis that occurs during the primary admission hospital stay during the first 7 days from randomization. Radiographic confirmation via CT imaging, ultrasound, duplex, transthoracic or trans-esophageal echo, or ventilation/perfusion scanning will be required. If an embolic event is unable to be verified radiographically, presumed or clinical suspicion of an embolic event will also be documented.
Acute respiratory distress syndrome (ARDS) in first 7 days | 7 days
  The Berlin definition for mild ARDS (PaO2/FIO2, ≤ 300 mmHg + timing, imaging and origin criteria) will be utilized as a threshold value to determine the incidence of ARDS
Abdominal compartment syndrome | Enrollment through hospital discharge or 28 days
  Intra-abdominal hypertension requiring paralysis, and/or diagnostic peritoneal lavage, and/or decompressive laparotomy
In-hospital mortality | Enrollment through hospital discharge or 28 days
  Death prior to hospital discharge
24-hour and 48-hour resuscitation | Enrollment through 24 hours and 48 hours
  All crystalloid, colloid (albumin) and plasma resuscitation, including the utilization of vitamin C
Acute kidney injury | Between 24 and 72 hours from the time of randomization
  At least one instance of a serum creatinine ≥ 1.5
Nosocomial Infection | 28 days
  CDC criteria for the diagnosis of hospital-acquired pneumonia and blood stream infection will be utilized
Ventilator-free days | 28 days
  Ventilator-free days will be determined by subtracting the number of ventilator days where mechanical ventilation was required utilizing an endotracheal tube or tracheostomy from 28 days. Patients undergoing operative interventions who remain on mechanical ventilation in the ICU will be considered to require ventilator support for that day.
ICU- free days | 28 days
  ICU-free days will be determined by subtracting the number of days where ICU admission was required from 28 days.
Allergic/transfusion reaction | Initial 12 hours from randomization
  Any transfusion complication during the initial 12 hours of enrollment will be documented. As the intervention is specific to the early phase of care setting and since transfusion complications are temporally related to the specific transfusion, transfusion-related complications will only be assessed during the initial 12 hours from randomization.
Persistent Organ Dysfunction (POD) Days | Starting at day of randomization and ending at day 28
  POD days will be determined based on the number of calendar days during which the patient was determined to be in POD (≥1 on total daily score), starting at day of randomization and ending at day 28.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Sperry, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with the funding agency as well as other researchers upon request to the Principal Investigator
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available after publication of the primary manuscript
Access Criteria: Requests for data will be submitted in writing and reviewed by the Principal Investigator.